CLINICAL TRIAL: NCT00631514
Title: Relevance of the Interaction Between Antihypertensive and Antirheumatic Drugs in a Family Practice
Brief Title: Interaction Between Antihypertensives and Non-Steroidal Anti-Inflammatory Drugs (NSAIDs)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Split (Other)
Collaborators: Dr Ivancica Pavlicevic Family Practice Office (Unknown)
Responsible Party: Ivancica Pavlicevic, Split University School of Medicine
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: 1-Pavlicevic
Record Dates: First submitted 2008-02-27; First posted 2008-03-07 (Estimated); Last update posted 2008-03-10 (Estimated); Status verified 2008-02

CONDITIONS: Hypertension
Keywords: antihypertensive drugs; non-steroidal anti-inflammatory drugs; interaction; family practice; arterial blood pressure
MeSH Terms: conditions — Hypertension | interventions — Acetaminophen; Ibuprofen; Piroxicam

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (No Intervention): Hypertensive persons taking either lisinopril/hydrochlorothiazide fixed combination or amlodipine all the time.
- 2 (Experimental): Intervention: NSAID. Hypertensives with osteoarthritis taking already amlodipine (5-10 mg o.d. per os) were randomized to the following drug interventions: to take either acetaminophen (1000 mg t.i.d. per os), piroxicam (10-20 mg o.d. per os) or ibuprofen (400-600 mg t.i.d. per os) for 1 month
  Interventions: Drug: acetaminophen; Drug: ibuprofen; Drug: piroxicam
- 3 (Experimental): Hypertensives with osteoarthritis taking already lisinopril/hydrochlorothiazide (20/12.5 mg o.d. per os), were sequentially randomized to the following drug interventions: acetaminophen (1000 mg t.i.d.), ibuprofen (400-600 mg t.i.d.) or piroxicam (10-20 mg o.d.), for 1 month each
  Interventions: Drug: acetaminophen; Drug: ibuprofen; Drug: piroxicam

INTERVENTIONS:
Drug: acetaminophen — acetaminophen 1000 mg t.i.d. per os ibuprofen 400-600 mg t.i.d. per os piroxicam 10-20 mg o.d. per os
  Other Names: paracetamol
  Arms: 2; 3
Drug: ibuprofen — acetaminophen 1000 mg t.i.d. per os ibuprofen 400-600 mg t.i.d. per os piroxicam 10-20 mg o.d. per os
  Arms: 2; 3
Drug: piroxicam — acetaminophen 1000 mg t.i.d. per os ibuprofen 400-600 mg t.i.d. per os piroxicam 10-20 mg o.d. per os
  Arms: 2; 3

SUMMARY:
NSAIDs may increase blood pressure and blunt the effects of many antihypertensives. Members of these drug classes differ in their propensity to such an interaction.

DETAILED DESCRIPTION:
To compare prospectively the effects of piroxicam, ibuprofen and acetaminophen on blood pressure control in hypertensive patients with osteoarthritis.

ELIGIBILITY:
Inclusion Criteria:

* Treated hypertensives of either gender aged between 55 and 76 years
* About 50% with concomitant osteoarthritis of the hip or knee

Exclusion Criteria:

* Normotensive persons or untreated hypertensives
* Individuals outside the age limits
* General exclusion criteria (e.g. uncooperative persons, advanced malignancies, participants in other studies)

Ages: 55 Years to 78 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2005-01; Primary Completion 2006-09 (Actual); Study Completion 2006-09 (Actual)

PRIMARY OUTCOMES:
Arterial blood pressure | 3 months (3 individual blocks of 1 month each)

SECONDARY OUTCOMES:
Body weight,serum electrolytes, urinary electrolytes (Na, K) | 3 months (3 periods of 1 month)

CONTACTS AND LOCATIONS:
Overall Officials: Zvonko - Rumboldt, MD, PhD, Study Director — Split University School of Medicine
Locations (1):
- Split University School of Medicine. Family Practice Department, Split, Croatia

REFERENCES:
- [Background] Pavlicevic I, Rumboldt M, Rumboldt Z. [Untoward interactions between antihypertensives and nonsteroidal anti-inflammatory drugs]. Lijec Vjesn. 2005 Jul-Aug;127(7-8):168-72. Croatian. PMID 16485829
- [Derived] Pavlicevic I, Kuzmanic M, Rumboldt M, Rumboldt Z. Interaction between antihypertensives and NSAIDs in primary care: a controlled trial. Can J Clin Pharmacol. 2008 Fall;15(3):e372-82. Epub 2008 Oct 24. PMID 18953082